CLINICAL TRIAL: NCT05526248
Title: A 2-stage, Lead-in and Randomized, Phase 2, Open-label Study of Darolutamide Versus Enzalutamide as Monotherapy on Testosterone Levels Change in Men With Hormone-Naïve Prostate Cancer
Brief Title: A Study Called ARAMON to Learn to What Extent Does Study Treatment With Darolutamide Affects Testosterone Levels in Men With Prostate Cancer That Had Not Been Treated With Hormonal Therapy Compared to Treatment With Enzalutamide
Acronym: ARAMON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21953
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Biochemically Recurrent Prostate Cancer
Keywords: Hormone-naive prostate cancer
MeSH Terms: interventions — darolutamide; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead-in phase: Darolutamide treatment (Experimental): Darolutamide treatment arm is single cohort in lead-in phase.
  Interventions: Drug: Darolutamide(BAY1841788, Nubeqa)
- Randomized phase: Darolutamide treatment (Experimental): The conduct of the randomized phase is dependent on the results of the lead-in phase.
  Interventions: Drug: Darolutamide(BAY1841788, Nubeqa)
- Randomized phase: Enzalutamide treatment (Active Comparator): The conduct of the randomized phase is dependent on the results of the lead-in phase.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Darolutamide(BAY1841788, Nubeqa) — tablet, oral
  Arms: Lead-in phase: Darolutamide treatment; Randomized phase: Darolutamide treatment
Drug: Enzalutamide — tablet, oral
  Arms: Randomized phase: Enzalutamide treatment

SUMMARY:
Researchers are looking for a better way to treat men who have biochemically recurrent hormone-naïve prostate cancer.

Hormone-naïve prostate cancer is a prostate cancer that has not yet been treated with hormonal therapy including androgen deprivation therapy (ADT). Biochemically recurrence (BCR) means that patients who received local treatment (surgery or radiation therapy) for prostate cancer now present with a rise in the blood level of a specific protein called PSA (prostate-specific antigen) but no detectable cancer or cancer spreading after a treatment that aimed to cure their prostate cancer (e.g. surgery and radiation). This may mean that the cancer has come back as the PSA level can be taken as a marker for prostate cancer development. Although men with BCR may not have symptoms for many years, proper treatment for BCR is important as the cancer may spread to other parts of the body in 7-8 years.

In prostate cancer patients, male sex hormones like testosterone (also called androgens) can sometimes help the cancer spread and grow. To reduce androgen levels in these patients, androgen deprivation therapy (ADT) is often used.

Second generation androgen receptor inhibitors including Darolutamide and Enzalutamide are available for the treatment of prostate cancer in addition to ADT. These inhibitors work by blocking androgen receptors and preventing it from attaching to proteins in cancer cells in the prostate. It is already known that men with prostate cancer benefit from these treatments. But besides benefits, Darolutamide and Enzalutamide are not without side effects.

Clinical studies have shown that treatment with Enzalutamide increase testosterone level in serum, probably because it can pass blood brain barrier and goes into the central nervous system (CNS). The increased testosterone levels are thought to cause some specific side effects including so called feminizing side effects like overdevelopment of the breast tissue in men, and breast tenderness. Darolutamide has a distinct chemical structure and reduced ability to enter the CNS compared with Enzalutamide. That means that Darolutamide potentially leads to fewer and less severe side effects than Enzalutamide.

In this study researchers will collect more data to learn to what extent Darolutamide affects serum testosterone levels in men with BCR in hormone-naïve prostate cancer. This study will consist of 2 stages. In stage 1 (also called lead-in phase) all participants will take Darolutamide by mouth twice a day. The study team will monitor and measure testosterone levels in the blood after:

* 12 weeks
* 24 weeks and
* 52 weeks of treatment.

The second stage (also called randomized phase) is conditional and depends on the results from the stage 1. It will be conducted if after 24 weeks of treatment with Darolutamide in stage 1:

* a mean change in blood testosterone levels is below 45% and
* if the feminizing side effects (including overdevelopment of the breast tissue in men, and breast tenderness) will occur less frequently than previously reported.

In the second stage of this study all participants will be randomly (by chance) assigned into two treatment groups, taking either Darolutamide twice daily or Enzalutamide once daily by mouth for a minimum of 12 and a maximum of 52 weeks.

During both stages of this study the study team will:

* do physical examinations
* take blood and urine samples
* examine heart health using ECG
* examine heart and lung health using CPET
* check bone density using x-ray scan (DEXA)
* check vital signs
* check if the participants' cancer has grown and/or spread using CT (computed tomography) or MRI (magnetic resonance imaging) and, if needed, bone scan
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

The study participants who receive Darolutamide in stage 2 can continue to receive their treatments as long as they benefit from the treatment. The participants from the Enzalutamide group can also switch to treatment with Darolutamide after finishing stage 2. The study team will continue to check the participants' health and collect information about medical problems that might be related to Darolutamide until up to 30 days of last dose for those participants who continue on treatment with Darolutamide.

ELIGIBILITY:
Inclusion Criteria:

* Male of ≥ 18 years of age.
* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate.
* Prior treatment with primary radical prostatectomy or definitive RT for localized prostate cancer
* Patients must have PSA ≥0.2 ng/mL after ART or SRT post-RP or after RP in participants who are unfit for ART or SRT, OR PSA ≥2 ng/mL above the nadir after primary RT only. (RP, radical prostatectomy; ART, adjuvant radiotherapy; SRT, salvage radiotherapy; RT primary radiotherapy)
* The presence of < 5 asymptomatic metastatic lesions on conventional or PSMA-PET based imaging methods permitted. Lesions that need treatment with any opioid based analgetic are considered symptomatic
* PSADT ≤ 20 months calculated per PCWG3 + RECIST 1.1 per Scher et al. (Scher et al. 2016) and MSKCC nomogram.
* Eastern Cooperative Oncology Group ECOG (PS) of 0 - 1.
* Serum testosterone >150 ng/dl.
* Patients must have adequate organ function within 4 weeks before the first dose of study intervention.
* More than 30 days (or 5 half-lives) (whichever is longer) since prior participation in another clinical trial with an investigational medicinal product.

Exclusion Criteria:

* Prior treatment with ADT of up to 6 months for localized disease is permitted but not if during the prior 6 months before first dose of study intervention. Plan to initiate ADT during the trial period is not allowed.
* Radiation therapy or major surgery within 4 weeks of screening.
* Systemic glucocorticoids within 3 months prior to the first dose or study intervention was expected to require systemic glucocorticoids during the study period
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association Class III or IV)
* Uncontrolled hypertension
* A gastrointestinal disorder or procedure which is expected to interfere significantly with absorption of study intervention.
* Prior history of a clinically significant malignancy with the exception of basal cell, squamous cell carcinoma of the skin, and superficial bladder cancer.
* Prior treatment with:

  * Second-generation androgen receptor (AR) inhibitors such as enzalutamide, apalutamide, darolutamide other investigational AR inhibitors
  * or Cytochrome P17 enzyme inhibitor such as abiraterone acetate as antineoplastic treatment for prostate cancer
* Prior history of gynecomastia
* Use of herbal products that may have had hormonal anti-prostate cancer activity or were known to decrease PSA levels (e.g., saw palmetto) within 4 weeks before the first dose of study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Unio Specialty Care - Urology - Sherman Oaks, Sherman Oaks, California
  - Mass General Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Oncology, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center New York - Main Campus, New York, New York
  - Central Ohio Urology Group - Gahanna, Gahanna, Ohio

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 participants were screened and signed the informed consent form for the study. Three participants were screen failures and did not complete screening. The study was conducted at five centers in the United States from 19 Dec 2022 (First Patient First Visit) to 4 Dec 2024 (Last Patient Last Visit). The randomized phase was never started based on the results of the lead-in phase.
Pre-assignment Details: Of the 25 who completed screening, 24 began the intervention, while one opted not to start.
Period: Overall Study
Arm/Group | Lead-in Phase: Darolutamide Treatment
Started (24) | 24
All Participants in the Lead-in Phase Had Been on Treatment for 12 Weeks | 24
Completed (20) | 20
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The evaluable set was defined as all enrolled participants having testosterone data at baseline and week 12. Enrolled participants include those who signed informed consent and met all inclusion and none of the exclusion criteria.
Arm/Group | Lead-in Phase: Darolutamide Treatment
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Number of participants with different baseline value of ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status scale is used to assess a patient's level of functioning and ability to carry out daily activities. Participants are staged based on their ECOG scores, which range from 0 to 5. In this framework, lower ECOG scores (0 and 1) indicate better outcomes, reflecting higher levels of functioning, while higher scores (3, 4, and 5) indicate worse outcomes, reflecting decreased levels of functioning and increased disability.
  Participants
    0 | 21
    1 | 2
Number of participants with different Gleason score of prostate cancer at initial diagnosis [Count of Participants; unit: Participants] — The Gleason score is a grading system used to evaluate the aggressiveness of prostate cancer based on the microscopic appearance of cancer cells. Participants are staged according to their Gleason scores, which typically range from 2 to 10. Lower Gleason scores (2-6) suggest better outcomes, reflecting less aggressive cancer, while higher scores (7-10) indicate worse outcomes, reflecting more aggressive and potentially harmful disease.
  Participants
    ≤ 6 | 6
    = 7 | 14
    ≥ 8 | 2
    Unknown | 1
Number of participants with Bone lesions at baseline [Count of Participants; unit: Participants]
  No | 18
  Yes | 5
Number of bone lesions at baseline [Count of Participants; unit: Participants] — Population: Of the 23 participants, only 5 presented bone lesions
  Participants
    number analyzed (Participants) | 5
    1 | 3
    4 | 2
Number of participants with different renal impairment [Count of Participants; unit: Participants]
  Normal: eGFR ≥ 90 mL/min | 6
  Mild impairment: 60 ≤ eGFR < 90 mL/min | 13
  Moderate impairment: 30 ≤ eGFR < 60 mL/min | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum Testosterone
Time Frame: From baseline to week 12
Population: The evaluable set was defined as all enrolled participants having testosterone data at baseline and week 12. Enrolled participants included those who signed informed consent and met all inclusion and none of the exclusion criteria.
Measure: Mean (95% Confidence Interval); unit: percentage (%)
Arm/Group | Lead-in Phase: Darolutamide Treatment
Number analyzed (Participants) | 22
percentage (%) | 53.46 [33.44 to 76.48]

2. Secondary Outcome: Percent Change in Serum Testosterone
Time Frame: From baseline to week 24 and 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage (%)
Arm/Group | Lead-in Phase: Darolutamide Treatment
Number analyzed (Participants) | 23
Percentage (%)
  Mean percent change from baseline at Week 24: number analyzed (Participants) | 21
  Mean percent change from baseline at Week 24 | 56.25 [39.87 to 74.55]
  Mean percent change from baseline at Week 52: number analyzed (Participants) | 20
  Mean percent change from baseline at Week 52 | 48.49 [32.76 to 66.08]

3. Secondary Outcome: Number of Participants With Different Serum Prostate-specific Antigen (PSA) Response
Description: PSA50 is defined as a ≥50% reduction of the PSA level compared to the baseline value, confirmed by a second subsequent PSA value with a ≥50% reduction from baseline 3 or more weeks later.
Time Frame: At week 4.12.24.36.52
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Darolutamide Treatment
Number analyzed (Participants) | 23
Participants
  Number of participants with confirmed PSA50 response at Week 4 | 23
  Number of participants with confirmed PSA50 response at Week 12 | 23
  Number of participants with confirmed PSA50 response at Week 24 | 23
  Number of participants with confirmed PSA50 response at Week 36 | 23
  Number of participants with confirmed PSA50 response at Week 52 | 23
  Number of participants with confirmed PSA50 response any time | 23

ADVERSE EVENTS:
Time Frame: Treatment-emergent AE (TEAE) was defined as any event arising or worsening after the first dose of study drug until 30 days after the last dose of study drug, up to 13 months.
Groups:
- Darolutamide 600 mg BID: Subjects received darolutamide 600 mg (BID) with food.
Arm/Group | Darolutamide 600 mg BID
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide 600 mg BID (N=24)
Retinal detachment (Eye disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide 600 mg BID (N=24)
Palpitations (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 7 (9)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 2 (2)
Anorectal infection (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (2)
Blood cholesterol increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Oestradiol increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (3)
Cardiac stress test abnormal (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Brain fog (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Libido decreased (Psychiatric disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 4 (4)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 19 (31)
Nipple pain (Reproductive system and breast disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Skin cyst excision (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 4 (7)
Hot flush (Vascular disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT05526248/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT05526248/SAP_001.pdf